CLINICAL TRIAL: NCT01989351
Title: LA PREDISPOSIZIONE AL DOLORE PERSISTENTE POST OPERATORIO IN AMBITO ORTOPEDICO: ASPETTI GENETICI
Brief Title: Predisposition to Persistent Pain After Orthopaedic Surgery: Genetic Aspects
Status: Completed | Type: Observational
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, Medical Doctor, ASST Gaetano Pini-CTO
Other Study IDs: IOGPGC03-13
Record Dates: First submitted 2013-11-05; First posted 2013-11-21 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VAS<4
- VAS>4

SUMMARY:
The study purpose is to examine polymorphism of genes associated to post-operative persistent pain and to verify the possible association between genotype phenotype and ADRB2 polymorphism in orthopaedic surgery. The primary aim is to evaluate the expression of ADBR2 in VAS>4 patients and to compare it to those with VAS<4.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* ASA I to III

Exclusion Criteria:

* Contraindications to regional anesthesia procedures
* Not stabilized neurological diseases
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total knee arthoplasty.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Frequency of SNPs rs12654788 and rs1042713 of ADBR2 gene in patients who complain persistent pain 4 months postoperatively compared to chronic pain free patients. | 4 months after surgery

SECONDARY OUTCOMES:
Expression frequency of OPRM1, COMT, IL1Ra | 6, 12, 24, 48 hours
Serum concentration of TNFα, TGFβ, IFNγ, IL-6 and IL-10 obtained with ELISA system | 6, 12, 24 and 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Cappelleri, MD, Principal Investigator — ASST Gaetano Pini-CTO; Manuela de Gregori, Biologist, Study Chair — Fondazione IRCCS Policlinico San Matteo di Pavia; Massimo Allegri, M.D., Study Chair — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (1):
- Istituto Ortopedico G. Pini, Milan, Milano, Italy